CLINICAL TRIAL: NCT03557697
Title: A Mobile Health Intervention to Reduce Diabetes Disparities in Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-00609; 5R00MD012811-05 (NIH)
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Type2 Diabetes
Keywords: Chinese Americans; SMS intervention
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wait-list control (Active Comparator): 3 measurement visits, baseline, 3, and 6 months
  Interventions: Behavioral: Standard of Care
- SMS intervention (Active Comparator): 3 measurement visits, baseline, 3, and 6 months
  Interventions: Behavioral: SMS Intervention

INTERVENTIONS:
Behavioral: Standard of Care — At the end of the study the control group will be provided with the opportunity to receive counseling videos delivered via SMS
  Arms: wait-list control
Behavioral: SMS Intervention — Participants in the intervention group will receive SMS based video counseling which include both educational and SCT=-based behavioral content. In addition, participants will receive biweekly phone calls from study community health workers to review the video content and clarify questions, set goals, and problem-solve barriers to achieving the goals.
  Arms: SMS intervention

SUMMARY:
Chinese Americans are one of the fastest growing immigrant groups in the US, who suffer disproportionately high type 2 diabetes (T2D) burden and have poorly controlled T2D. Despite the well-documented T2D disparities in this minority group, limited work has been conducted to improve health outcomes in Chinese Americans. The goal of this Pathway to Independence Award (K99/R00) is to expedite the candidate's transition to an independent investigator who possesses focused expertise in development and evaluation of culturally and linguistically tailored and sustainable interventions to reduce T2D disparities in Chinese Americans. In the K99 phase of this award, the candidate will obtain critical training needed to accomplish this goal and will develop a short message service (SMS) intervention to improve T2D management in Chinese Americans.

More specifically, the aims are to 1) characterize barriers and facilitators of glycemic control in Chinese Americans with T2D (Aim 1a); 2) develop culturally and linguistically tailored SMS intervention content (Aim 1b); and 3) assess the feasibility and acceptability of the SMS intervention in a pre-, post-test study (Aim 1c).

In the R00 phase, the candidate will refine the SMS intervention based on the K99 pilot data and evaluate the proof-of-concept regarding its efficacy in a pilot randomized controlled trial among 66 Chinese Americans with T2D (Aim 2). Participants will be randomized to one of 2 arms (n=30 each): 1) wait-list control and 2) SMS intervention. Both groups will continue to receive standard of care treatment for their T2D. The SMS group will receive brief lifestyle counseling videos via SMS links. At the end of the study, the wait-list control group will be provided the opportunity to receive the SMS-based counseling videos. Measurements will be obtained at baseline, 3, and 6 months. The primary outcome is HbA1c and secondary outcomes include self-efficacy, diabetes self-management behaviors, dietary intake and physical activity behaviors. Linear mixed modeling will be used to examine the group and group by time interaction effects between the SMS intervention and wait-list control group. Findings from this R00 study will inform a larger full-scale R01 efficacy trial of the SMS intervention, and ultimately, establish the candidate's program of research focused on developing and testing sustainable interventions to reduce disparities in chronic disease outcomes in Chinese Americans. This project can serve as a program model for other chronic disease interventions in Chinese Americans that require lifestyle modification (e.g., prediabetes, hypertension), or for disparities research in other high-risk immigrant populations (e.g., South Asians, Hispanic Americans).

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Chinese Immigrant or Chinese American
* be able to speak and understand Mandarin
* self-report a diagnosis of T2D
* baseline HbA1c ≥ 7%
* be currently using WeChat or text messages• be willing to receive WeChat or text messages regarding T2D management
* express strong interest and confidence in finishing watching 2 diabetes videos each week for a total of 12 weeks
* express motivation to make lifestyle changes to control their diabetes
* be willing to wear ActiGraph for 8 days

Exclusion Criteria:

* unable or unwilling to provide informed consent
* unable to participate meaningfully in the intervention (e.g., uncorrected sight and hearing impairment)
* unwilling to accept randomization assignment
* pregnant, plans to becomes pregnant in the next 6 months, or who become pregnant during the study
* breastfeeding
* live in a facility or other health care setting where they have to control over diabetes self-management

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hu, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Requests should be directed to Lu.Hu@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Liu J, Cao J, Shi Y, Sevick MA, Islam N, Feldman N, Li H, Wang C, Zhao Y, Tamura K, Levy N, Jiang N, Zhu Z, Wang Y, Hong J, Hu L. A Culturally and Linguistically Tailored Intervention to Improve Diabetes-Related Outcomes in Chinese Americans With Type 2 Diabetes: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Oct 27;13:e78036. doi: 10.2196/78036. PMID 41144955
- [Derived] Shi Y, Sevick MA, Tang H, Wang C, Zhao Y, Yoon S, Li H, Jiang Y, Bai Y, Ong IH, Yang X, Su L, Levy N, Tamura K, Hu L. Culturally Tailored Social Media Intervention Improves Health Outcomes in Chinese Americans with Type 2 Diabetes: Preliminary Evidence from a Pilot RCT. J Gen Intern Med. 2025 Jul;40(10):2319-2329. doi: 10.1007/s11606-025-09430-9. Epub 2025 Feb 27. PMID 40016380
- [Derived] Hu L, Islam N, Zhang Y, Shi Y, Li H, Wang C, Sevick MA. Leveraging Social Media to Increase Access to an Evidence-Based Diabetes Intervention Among Low-Income Chinese Immigrants: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Oct 28;11(10):e42554. doi: 10.2196/42554. PMID 36306161

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wait-list Control | SMS Intervention
Started | 30 | 30
Completed | 28 | 26
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait-list Control | SMS Intervention | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (11.4) | 55.6 (11.5) | 54.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Plasma Glucose Concentration Measured by Hemoglobin A1c (HbA1c) Levels
Description: HbA1c testing results abstracted from medical record.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Percentage | -0.68 [-1.14 to -0.22] | -0.95 [-1.45 to -0.46]

2. Primary Outcome: Change in Average Plasma Glucose Concentration Measured by Hemoglobin A1c (HbA1c) Levels
Description: HbA1c testing results abstracted from medical record.
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Percentage | -0.82 [-1.30 to -0.34] | -1.08 [-1.58 to -0.58]

3. Secondary Outcome: Change in Stanford Diabetes Self-Efficacy Scale Score
Description: 8-item questionnaire asking participants to rate their confidence level in performing specific Type 2 Diabetes self-management behaviors on 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident). The total score is the sum of responses and ranges from 8-80; higher scores indicate higher levels of confidence in performing self-management behaviors.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | -2.72 [-6.93 to 1.50] | 5.76 [1.45 to 10.06]

4. Secondary Outcome: Change in Stanford Diabetes Self-Efficacy Scale Score
Description: as for outcome 3
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.21 [-4.07 to 4.48] | 6.08 [1.72 to 10.44]

5. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - General Diet Score
Description: The SDSCA measures the frequency of diabetes self-care activities over the previous week across five domains of self-care. The General Diet subscale comprises 2 items rated on a scale from 0-7. The total General Diet score is the mean of the item responses and ranges from 0-14, with higher scores indicating better compliance.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.43 [-0.37 to 1.23] | 2.04 [1.21 to 2.86]

6. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - General Diet Score
Description: as for outcome 5
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.09 [-0.72 to 0.91] | 1.74 [0.90 to 2.57]

7. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Specific Diet Score
Description: The SDSCA measures the frequency of diabetes self-care activities over the previous week across five domains of self-care. The Specific Diet subscale comprises 2 items rated on a scale from 0-7. The total Specific Diet score is the mean of the item responses and ranges from 0-14, with higher scores indicating better compliance.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | -0.31 [-0.93 to 0.32] | 0.17 [-0.47 to 0.81]

8. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Specific Diet Score
Description: as for outcome 7
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.2 [-0.43 to 0.84] | 0.59 [-0.06 to 1.24]

9. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Exercise Score
Description: The SDSCA measures the frequency of diabetes self-care activities over the previous week across five domains of self-care. The Exercise subscale comprises 2 items rated on a scale from 0-7. The total Exercise score is the mean of the item responses and ranges from 0-14, with higher scores indicating better compliance.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.20 [-0.61 to 1.01] | 1.26 [0.43 to 2.10]

10. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Exercise Score
Description: as for outcome 9
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.89 [0.07 to 1.72] | 1.56 [0.71 to 2.40]

11. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Blood-Glucose Testing Score
Description: The SDSCA measures the frequency of diabetes self-care activities over the previous week across five domains of self-care. The Blood-Glucose Testing subscale comprises 2 items rated on a scale from 0-7. The total Blood-Glucose Testing score is the mean of the item responses and ranges from 0-14, with higher scores indicating better compliance.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | -0.70 [-1.68 to 0.28] | 0.47 [-0.52 to 1.46]

12. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Blood-Glucose Testing Score
Description: as for outcome 11
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | -0.14 [-1.13 to 0.86] | 0.10 [-0.90 to 1.11]

13. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Foot Care Score
Description: The SDSCA measures the frequency of diabetes self-care activities over the previous week across five domains of self-care. The Foot Care subscale comprises 2 items rated on a scale from 0-7. The total Foot Care score is the mean of the item responses and ranges from 0-14, with higher scores indicating better compliance.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.00 [-0.63 to 0.63] | -0.22 [-0.88 to 0.44]

14. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Foot Care Score
Description: as for outcome 13
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | -0.17 [-0.81 to 0.47] | 0.07 [-0.60 to 0.73]

15. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Medication Adherence Score
Description: The SDSCA measures the frequency of diabetes self-care activities over the previous week across five domains of self-care. The Medication Adherence subscale comprises 3 items rated on a scale from 0-7. The total Medication Adherence score is the mean of the item responses and ranges from 0-21, with higher scores indicating better compliance.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.06 [-0.49 to 0.62] | -0.03 [-0.59 to 0.53]

16. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) - Medication Adherence Score
Description: as for outcome 15
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | -0.06 [-0.63 to 0.51] | -0.46 [-1.03 to 0.11]

17. Secondary Outcome: Change in Starting The Conversation Scale: Fruits
Description: The Starting The Conversation Scale contains 6 items and asks respondents about the types of food they consumed in the past 30 days. The Fruit subscale comprises 1 item in which respondents indicate how many cups of fruit, on average, they ate each day in the past 30 days. The total score is estimation of average cups of fruit consumed per day.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.44 [-0.74 to -0.13] | 0.15 [-0.15 to 0.46]

18. Secondary Outcome: Change in Starting The Conversation Scale: Fruits
Description: The Starting The Conversation Scale contains 6 items and asks respondents about the types of food they consumed in the past 30 days. The Fruit subscale comprises 1 item in which respondents indicate how many cups of fruits, on average, they ate each day in the past 30 days. The total score is estimation of average cups of fruit consumed per day.
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.32 [-0.63 to -0.01] | 0.17 [-0.14 to 0.48]

19. Secondary Outcome: Change in Starting The Conversation Scale: Vegetables
Description: The Starting The Conversation Scale contains 6 items and asks respondents about the types of food they consumed in the past 30 days. The Vegetables subscale comprises 1 item in which respondents indicate how many cups of vegetables, on average, they ate each day in the past 30 days. The total score is estimation of average cups of vegetables consumed per day.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.06 [-0.49 to 0.37] | 0.22 [-0.22 to 0.65]

20. Secondary Outcome: Change in Starting The Conversation Scale: Vegetables
Description: as for outcome 19
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | 0.00 [-0.43 to 0.43] | 0.52 [0.07 to 0.96]

21. Secondary Outcome: Change in Starting The Conversation Scale: Refined Grains
Description: The Starting The Conversation Scale contains 6 items and asks respondents about the types of food they consumed in the past 30 days. The Refined Grains subscale comprises 1 item in which respondents indicate how many cups of refined grains, on average, they ate each day in the past 30 days. The total score is estimation of average cups of refined grains consumed per day.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.20 [-0.54 to 0.14] | -0.59 [-0.93 to -0.24]

22. Secondary Outcome: Change in Starting The Conversation Scale: Refined Grains
Description: as for outcome 21
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.20 [-0.54 to 0.15] | -0.34 [-0.70 to 0.01]

23. Secondary Outcome: Change in Starting The Conversation Scale: Whole Wheat
Description: The Starting The Conversation Scale contains 6 items and asks respondents about the types of food they consumed in the past 30 days. The Whole Wheat subscale comprises 1 item in which respondents indicate how many cups of whole wheat, on average, they ate each day in the past 30 days. The total score is estimation of average cups of whole wheat consumed per day.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.18 [-0.47 to 0.11] | -0.12 [-0.42 to 0.18]

24. Secondary Outcome: Change in Starting The Conversation Scale: Whole Wheat
Description: as for outcome 23
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.03 [-0.33 to 0.27] | 0.08 [-0.23 to 0.38]

25. Secondary Outcome: Change in Starting The Conversation Scale: Sugary Drinks
Description: The Starting The Conversation Scale contains 6 items and asks respondents about the types of food they consumed in the past 30 days. The Sugary Drinks subscale comprises 1 item in which respondents indicate how many cans of sugary drinks, on average, they consumed each day in the past 30 days. The total score is estimation of average cans of sugary drinks consumed per day.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: Cans/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cans/day | -0.10 [-0.25 to 0.04] | -0.16 [-0.31 to -0.01]

26. Secondary Outcome: Change in Starting The Conversation Scale: Sugary Drinks
Description: as for outcome 25
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Cans/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cans/day | -0.01 [-0.15 to 0.14] | -0.1 [-0.25 to 0.05]

27. Secondary Outcome: Change in Starting The Conversation Scale: Starchy Foods
Description: The Starting The Conversation Scale contains 6 items and asks respondents about the types of food they consumed in the past 30 days. The Starchy Foods subscale comprises 1 item in which respondents indicate how many cups of starchy foods, on average, they ate each day in the past 30 days. The total score is estimation of average cups of starchy foods consumed per day.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.07 [-0.32 to 0.18] | -0.24 [-0.50 to 0.02]

28. Secondary Outcome: Change in Starting The Conversation Scale: Starchy Foods
Description: as for outcome 27
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Cups/day
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
Cups/day | -0.1 [-0.35 to 0.16] | -0.33 [-0.59 to -0.07]

29. Secondary Outcome: Change in International Physical Activity Questionnaire (IPAQ) Score
Description: 7-item self-assessment providing an estimate of the number of minutes per week participants engage in three categories of physical activity: vigorous activity, moderate activity, and walking activity. Results are expressed in metabolic equivalent (MET) minutes per week. MET minutes represent the amount of energy expended carrying out physical activity. Higher scores indicate higher weekly levels of physical activity.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: metabolic equivalent (MET) minutes/week
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
metabolic equivalent (MET) minutes/week | 25.58 [-949.66 to 1000.81] | -196.14 [-1195.91 to 803.64]

30. Secondary Outcome: Change in International Physical Activity Questionnaire (IPAQ) Score
Description: as for outcome 29
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: metabolic equivalent (MET) minutes/week
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
metabolic equivalent (MET) minutes/week | 1032.79 [46.2 to 2019.38] | 199.57 [-812.43 to 1211.56]

31. Secondary Outcome: Change in Belief in Self-Management Score
Description: Participants rated the importance of five self-care behaviors related to diabetes self-care-following a diabetic diet, exercising, self-monitoring blood glucose, taking medication, and checking their feet. Each behavior was rated on a 5-point Likert scale, where 1 indicated "not important" and 5 indicated "very important." The total score is calculated as the mean of the item responses and ranges from 1-5, with higher scores indicating greater belief in the importance of diabetes self-management.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.21 [0.02 to 0.40] | 0.05 [-0.15 to 0.24]

32. Secondary Outcome: Change in Belief in Self-Management Score
Description: as for outcome 31
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.21 [0.02 to 0.40] | 0.14 [-0.06 to 0.34]

33. Secondary Outcome: Change in Diabetes Distress Scale Score
Description: This 17-item scale required participants to rate the extent to which each item was problematic for them in the past month, using a 6-point Likert scale ranging from 1 (no problem) to 6 (serious problem). The total score is the mean of the item scores and ranges from 1-6, with higher scores indicating a greater level of distress.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.01 [-0.18 to 0.20] | -0.24 [-0.44 to -0.04]

34. Secondary Outcome: Change in Diabetes Distress Scale Score
Description: as for outcome 33
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control | SMS Intervention
Number analyzed (Participants) | 30 | 30
score on a scale | 0.06 [-0.13 to 0.25] | -0.37 [-0.58 to -0.17]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Wait-list Control | SMS Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03557697/Prot_SAP_000.pdf